CLINICAL TRIAL: NCT02664922
Title: Anesthetic Techniques and the Effect on Cardiac Electrophysiology Procedures
Brief Title: Anesthetic Techniques in EP Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor study design and too many study groups.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Anes Tech 11-003514
Record Dates: First submitted 2014-10-05; First posted 2016-01-27 (Estimated); Results first posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Cardiac Disease
Keywords: Electrophysiology; Anesthetics
MeSH Terms: conditions — Heart Diseases | interventions — Propofol; Ketamine; Remifentanil; Sevoflurane

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sedation - Group 1 (Experimental): Sedation - monitored anesthesia with propofol.
  Interventions: Drug: Propofol
- Sedation - Group 2 (Experimental): Sedation - monitored anesthesia with ketamine + propofol
  Interventions: Drug: Propofol; Drug: Ketamine
- Sedation - Group 3 (Experimental): Sedation - monitored anesthesia with remifentanil + propofol
  Interventions: Drug: Propofol; Drug: Remifentanil
- General Anesthesia - Group 1 (Experimental): General anesthesia (GA) with Sevoflurane + O2
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — 1 of 3 sedation groups for SVT, RVOT/PVC ablation, and aflutter procedures.
  1 of 2 sedation groups for VT ablation and afib procedures.
  Other Names: Diprivan
  Arms: Sedation - Group 1; Sedation - Group 2; Sedation - Group 3
Drug: Ketamine — 1 of 3 sedation groups for SVT, RVOT/PVC ablation, and aflutter procedures.
  1 of 2 sedation groups for VT ablation and afib procedures.
  Other Names: Ketalar
  Arms: Sedation - Group 2
Drug: Remifentanil — 1 of 3 sedation groups for SVT, RVOT/PVC ablation, and aflutter procedures.
  Other Names: Ultiva
  Arms: Sedation - Group 3
Drug: Sevoflurane — 1 general anesthesia group for VT ablations and afib procedures.
  Other Names: Ultane
  Arms: General Anesthesia - Group 1

SUMMARY:
The purpose of this study is to compare different combinations of anesthetic drugs (cause loss of sensation) in terms of effectiveness, adverse effects, pain relief, and patient comfort for cardiac electrophysiology procedures. In addition, the investigators are studying the different anesthetic combinations to determine the best approach in terms of identification and treatment of arrhythmias.

DETAILED DESCRIPTION:
Anesthetic management in patients coming for electrophysiology procedures is extremely important and hemodynamically challenging in order to minimize interference on the electrophysiology studies (EPS) and the ability to trigger arrhythmias while also maintaining patient comfort and limited movement. Various anesthetic combinations are administered to provide sedation, analgesia/sedation, or general anesthesia. The ideal agent should produce rapid loss of consciousness while ensuring cardiovascular stability and prompt recovery with few adverse effects. Our goal is to study anesthetic techniques and the effect on electrophysiology procedures to determine the best anesthetic combination in terms of effectiveness, adverse effects, pain relief, and patient comfort.

Adult patients scheduled for electrophysiology procedures will be enrolled in the study and randomly assigned to an anesthetic group based on their schedule procedure. Sedation cases for supraventricular tachycardia (SVT), right ventricular outflow tract (RVOT)/premature ventricular contraction (PVC) ablation, and atrial flutter (aflutter) procedures will be randomly assigned to one of three groups: 1) monitored anesthesia (local anesthesia with sedation and analgesia/pain reliever) with propofol (induce sleep), 2) monitored anesthesia with ketamine (sedation) + propofol (induce sleep), or 3) monitored anesthesia with remifentanil infusion (pain reliever) + propofol (induce sleep). Sedation cases for ventricular tachycardia (VT) ablation and atrial fibrillation (afib) procedures will be randomly assigned to one of two groups: 1) monitored anesthesia (local anesthesia with sedation and analgesia/pain reliever) with propofol (induce sleep), or 2) monitored anesthesia with ketamine (sedation) + propofol (induce sleep). General anesthesia (GA) cases, including VT ablation and afib procedures will receive general anesthesia (state of unconsciousness) with sevoflurane (loss of consciousness) + O2. Anesthesia factors, such as hemodynamics and cerebral oxygen saturation will be continuously monitored and recorded throughout the study. In addition, we will be looking at standard echocardiogram and electrophysiology (EP) parameters. The patient's pain level, level of sedation, and satisfaction will also be measured using scales, assessments, and surveys.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for cardiac electrophysiology procedures
* Patients ≥18 years of age

Exclusion Criteria:

* Gastroesophageal reflux disease (GERD),
* pulmonary hypertension,
* severe pulmonary disease,
* obstructive sleep apnea (OSA) with continuous positive airway pressure therapy (CPAP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2012-05 (Actual); Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aman Mahajan, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ronald Reagan UCLA Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sedation - Group 1: Sedation - monitored anesthesia with propofol.
  Propofol: 1 of 3 sedation groups for SVT, RVOT/PVC ablation, and aflutter procedures.
  1 of 2 sedation groups for VT ablation and afib procedures.
- Sedation - Group 2: Sedation - monitored anesthesia with ketamine + propofol
  Propofol: 1 of 3 sedation groups for SVT, RVOT/PVC ablation, and aflutter procedures.
  1 of 2 sedation groups for VT ablation and afib procedures.
  Ketamine: 1 of 3 sedation groups for SVT, RVOT/PVC ablation, and aflutter procedures.
  1 of 2 sedation groups for VT ablation and afib procedures.
- Sedation - Group 3: Sedation - monitored anesthesia with remifentanil + propofol
  Propofol: 1 of 3 sedation groups for SVT, RVOT/PVC ablation, and aflutter procedures.
  1 of 2 sedation groups for VT ablation and afib procedures.
  Remifentanil: 1 of 3 sedation groups for SVT, RVOT/PVC ablation, and aflutter procedures.
Period: Overall Study
Arm/Group | Sedation - Group 1 | Sedation - Group 2 | Sedation - Group 3 | General Anesthesia - Group 1
Started | 11 | 12 | 7 | 5
Completed | 10 | 12 | 7 | 5
Not Completed | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sedation - Group 1 | Sedation - Group 2 | Sedation - Group 3 | General Anesthesia - Group 1 | Total
Number analyzed (Participants) | 10 | 12 | 7 | 5 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (16) | 56 (13) | 48 (18) | 43 (16) | 53 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 2 | 1 | 13
  Male | 4 | 8 | 5 | 4 | 21

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Anesthetic Drugs in Terms of Number of Participants With Adverse Events.
Description: Direct observation and medical record review will be used to analyze adverse effects. Reported as number of participants with one or more adverse events.
Time Frame: Intraoperatively to postoperatively in the ICU, an expected average of 5-7 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | Sedation - Group 1 | Sedation - Group 2 | Sedation - Group 3 | General Anesthesia - Group 1
Number analyzed (Participants) | 10 | 12 | 7 | 5
Participants | 1 | 2 | 0 | 0

2. Primary Outcome: Effectiveness of Anesthetic Drugs in Terms of Pain Relief.
Description: A patient's pain level will be assessed using a numerical pain rating scale from 0 "no pain" to 10 "worst possible pain".
Time Frame: Intraoperatively to postoperatively in the ICU, an expected average of 5-7 hours.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedation - Group 1 | Sedation - Group 2 | Sedation - Group 3 | General Anesthesia - Group 1
Number analyzed (Participants) | 10 | 12 | 7 | 5
score on a scale | 1.7 (1.3) | 0.4 (0.5) | 0.2 (0.5) | 0 (0)

3. Primary Outcome: Effectiveness of Anesthetic Drugs in Terms of Patient Comfort.
Description: A patient's level of sedation will be assessed using a scoring system on a scale from 1-5. The Observer's Assessment of Alertness/Sedation (OAA/S) Score Responsiveness Component score from 1 - Does not respond to mild prodding or shaking to 5 - Responds readily to name spoken in normal tone.
Time Frame: Intraoperatively to postoperatively in the ICU, an expected average of 5-7 hours.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedation - Group 1 | Sedation - Group 2 | Sedation - Group 3 | General Anesthesia - Group 1
Number analyzed (Participants) | 10 | 12 | 7 | 5
score on a scale | 2.9 (1.2) | 3.0 (1.3) | 3.0 (1.3) | 1.0 (0.0)

4. Primary Outcome: Effectiveness of Anesthetic Drugs in Terms of Patient Satisfaction.
Description: Patients will also be asked to complete a written questionnaire prior to discharge from the hospital to measure patient satisfaction during their anesthesia care. A Likert Scale is used and ranges from 1 - Disagree very much to 6 - Agree very much.
Time Frame: Intraoperatively to postoperatively in the ICU, an expected average of 5-7 hours.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedation - Group 1 | Sedation - Group 2 | Sedation - Group 3 | General Anesthesia - Group 1
Number analyzed (Participants) | 10 | 12 | 7 | 5
score on a scale | 3.4 (0.4) | 3.0 (0.7) | 3.5 (0.5) | 3.1 (0.1)

5. Secondary Outcome: Effectiveness of Anesthetic Drugs in Terms of Proceduralist Satisfaction.
Description: The proceduralist will complete a written questionnaire after the procedure to rate their satisfaction. A Likert Scale is used and ranges from 1 - Disagree very much to 6 - Agree very much.
Time Frame: Intraoperatively to postoperatively in the ICU, an expected average of 5-7 hours.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sedation - Group 1 | Sedation - Group 2 | Sedation - Group 3 | General Anesthesia - Group 1
Number analyzed (Participants) | 10 | 12 | 7 | 5
score on a scale | 5.7 (0.4) | 5.6 (0.5) | 5.2 (0.3) | 5.1 (1.9)

6. Secondary Outcome: Effectiveness of Anesthetic Drugs in Terms of Number of Participants With Clinical Success.
Description: The proceduralist will follow-up 1-3 months post-procedure to evaluate the number of participants with clinical success reported by number of recurrences. Clinical success is defined as 0 recurrences in participants at 1-3 months post-operatively.
Time Frame: 1-3 months postoperatively
Population: Patients were excluded from analysis if there was no electrophysiology follow-up in the medical record 1-3 months postoperatively.
Measure: Count of Participants; unit: Participants
Arm/Group | Sedation - Group 1 | Sedation - Group 2 | Sedation - Group 3 | General Anesthesia - Group 1
Number analyzed (Participants) | 3 | 5 | 3 | 4
Participants | 0 | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Intraoperatively to postoperatively in the ICU, an expected average of 5-7 hours, and up to 5 days.
Arm/Group | Sedation - Group 1 | Sedation - Group 2 | Sedation - Group 3 | General Anesthesia - Group 1
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/7 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/10 | 2/12 | 0/7 | 1/5
Other Adverse Events (participants affected / at risk) | 1/10 | 2/12 | 0/7 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedation - Group 1 (N=10) | Sedation - Group 2 (N=12) | Sedation - Group 3 (N=7) | General Anesthesia - Group 1 (N=5)
New onset atrial fibrillation requiring cardioversion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 | 1 (1)
VA ECMO (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiorgan Failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Death (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sedation - Group 1 (N=10) | Sedation - Group 2 (N=12) | Sedation - Group 3 (N=7) | General Anesthesia - Group 1 (N=5)
slow ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
non-sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial Drain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes